CLINICAL TRIAL: NCT00327938
Title: Genetically Variation - May the Need of Opioids During Surgery be Known Beforehand by Giving Noxious Stimulation and Measure the Skin Conductance Response Before Surgery?
Brief Title: Genetic Variation - The Need for Opioids During Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rikshospitalet University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2.2005.2354
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Pain
Keywords: Remifentanil; Skin Conductance; Anesthesia; Analgesics, Opioid
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Measuring of skin conductance
Procedure: Tetanic stimuli

SUMMARY:
The purpose of this study is to find out if the tetanic noxious stimuli and the measured skin conductance response can be used as a test in patients before surgery to have an indication about what amount of analgesics the patient will need during surgery.

DETAILED DESCRIPTION:
Skin Conductance (SC) shows the emotional state as reflected in changes in the sympathetic nervous system. During sleep or other states of low basic sympathetic activity, activation of the sympathetic nervous system results in filling of the palmar and plantar sweat glands, and the SC increases transiently before the sweat is removed and the SC decreases again. When a short lasting outgoing sympathetic nervous burst occurs, fluctuations of SC will follow. An increase in the number of SC fluctuations (NSCF) can therefore be interpreted as increased activity in this part of the sympathetic nervous system. When remifentanil, an opioid analgetic is given, NSCF is reduced.

Genetic variation influences the pharmacokinetics and the pharmacodynamics of analgesics like morphine derivates and remifentanil. 50 female patients will therefore be blood tested to study if they are Val/Val or Met/Met for the COMT gene, or if they are homozygous or heterozygous for the 118G allele and the 118A allele.

This study will show if skin conductance can be used to measure noxious stimulation response before surgery (by giving a tetanic stimuli), and then predict what level of analgesic a patient will need during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women in American Society of Anesthesiologists (ASA) group 1-2 and with body mass index between 20 and 30 and going through laparoscopic surgery at the Gynecological Department, Ullevål University Hospital.
* Normal renal and hepar function (serum albumin and serum creatinine should be within the normal limit).

Exclusion Criteria:

* Chronic pain in the last 6 months or recent use and abuse of analgesics.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2006-05

PRIMARY OUTCOMES:
skin conductance response

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Storm, PhD, Study Director — Rikshospitalet University Hospital
Locations (1):
- Ulleval University Hospital, Oslo, Norway